CLINICAL TRIAL: NCT03396861
Title: Subconjunctival Aflibercept Injection for Pseudophakic Cystoid Macular Edema
Brief Title: Treatment of Macular Edema After Cataract Surgery with Subconjunctival Aflibercept
Acronym: ACME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Tufts Medical Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12338
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Irvine-Gass Syndrome
Keywords: macular edema; pseudophakia; pseudophakic macular edema; retinal swelling; aflibercept; anti-vascular endothelial growth factor; subconjunctival injection
MeSH Terms: conditions — Macular Edema; Pseudophakia | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subconjunctival aflibercept (Experimental): Subconjunctival aflibercept 2 milligrams (mg) /0.05 milliliters (mL) administered at baseline visit and possibly again at Month 1 visit depending on initial response.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Subconjunctival aflibercept

SUMMARY:
This research study is being conducted to determine the safety and tolerability of subconjunctival injections of aflibercept in the treatment of pseudophakic cystoid macular edema that has not responded well to first-line standard of care treatment (eye drops).

Pseudophakic cystoid macular edema (CME) is swelling of the retina that can occur weeks or years after cataract surgery and typically results in decreased vision. Subconjunctival injections are injections placed just beneath the clear membrane (conjunctiva) of the eye.

A recent report of one patient who received two subconjunctival injections of a similar medication to the one being studied here indicated that subconjunctival injections of this class of medication may be an effective and less invasive alternative to intravitreal injections for pseudophakic CME. Because of the similarity of the drugs and the patient's treatment success, we would like to see if subconjunctival injection(s) of aflibercept will work in treating pseudophakic CME. If successful, the risk of an intraocular infection and glaucoma that comes with standard of care treatments might be greatly reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with pseudophakic CME defined as central retinal thickness (CRT)>300 microns, presence of intraretinal cysts on optical coherence tomography (OCT) and visual acuity <=20/32 with petaloid leakage on fluorescein angiogram and late leakage at the disc
2. Diagnosed with "recalcitrant" CME, defined as less than a 15% decrease in CRT after at least 6 weeks of topical non-steroidal anti-inflammatory drug
3. Has had cataract surgery in the study eye with posterior chamber or anterior chamber intraocular lens implantation
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent

Exclusion Criteria:

1. Retinal diseases (including diabetic retinopathy, retinal vein or artery occlusion, neovascular age-related macular degeneration, radiation retinopathy, vitreomacular traction, epiretinal membrane).
2. Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye.
3. Active infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye.
4. Prior treatment with sub-Tenon's or intravitreal steroids.
5. Prior treatment with an intravitreal anti-vascular endothelial growth factor (VEGF) agent in the study eye or systemic administration of anti-VEGF.
6. Use of topical prostaglandin analogues or pilocarpine.
7. Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with glaucoma medications.
8. Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye.
9. Vision loss in the study eye, determined by the investigator to be from a cause other than CME, e.g. optic neuropathy, end-stage glaucoma.
10. Any significant media opacity including vitreous hemorrhage or corneal scarring.
11. Fluorescein dye allergy or intolerance
12. Allergy to aflibercept or any of the components
13. Cerebrovascular accident or myocardial infarction within 1 year of the screening visit.
14. Pregnant or breast-feeding women
15. Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception starting at least 2 menstrual cycles prior to the baseline visit, during the study and in the 3 months immediately following the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Month 2
  Systemic and ocular adverse events of subconjunctivally administered aflibercept injection in the treatment of pseudophakic cystoid macular edema at Month 2

SECONDARY OUTCOMES:
Change in visual acuity | Month 2 and Month 6
  Change in best-corrected visual acuity at Months 2 and 6
Change in central retinal thickness | Month 2 and Month 6
  Change in central retinal thickness as measured by optical coherence tomography at Months 2 and 6
Proportion of patients needing re-treatment | Month 1
  Proportion of patients needing subconjunctival aflibercept injection treatment at Month 1
Proportion of patients needing additional non-study treatment though Month 6 | Month 6
  Proportion of patients receiving additional non-study treatment (e.g. periocular or intravitreal steroid) through Month 6
Adverse Events - end of study period | Month 6
  Incidence and severity of systemic and ocular events at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Elias Reichel, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muakkassa NW, Klein KA, Hamrah P, Reichel E. Subconjunctival Bevacizumab for the Treatment of Keratoprosthesis-Associated Cystoid Macular Edema. Ophthalmic Surg Lasers Imaging Retina. 2016 Mar;47(3):276-9. doi: 10.3928/23258160-20160229-11. PMID 26985802
- [Background] Guo S, Patel S, Baumrind B, Johnson K, Levinsohn D, Marcus E, Tannen B, Roy M, Bhagat N, Zarbin M. Management of pseudophakic cystoid macular edema. Surv Ophthalmol. 2015 Mar-Apr;60(2):123-37. doi: 10.1016/j.survophthal.2014.08.005. Epub 2014 Sep 2. PMID 25438734
- [Background] Arevalo JF, Garcia-Amaris RA, Roca JA, Sanchez JG, Wu L, Berrocal MH, Maia M; Pan-American Collaborative Retina Study Group. Primary intravitreal bevacizumab for the management of pseudophakic cystoid macular edema: pilot study of the Pan-American Collaborative Retina Study Group. J Cataract Refract Surg. 2007 Dec;33(12):2098-105. doi: 10.1016/j.jcrs.2007.07.046. PMID 18053911
- [Background] Lin CJ, Tsai YY. USE OF AFLIBERCEPT FOR THE MANAGEMENT OF REFRACTORY PSEUDOPHAKIC MACULAR EDEMA IN IRVINE-GASS SYNDROME AND LITERATURE REVIEW. Retin Cases Brief Rep. 2018 Winter;12(1):59-62. doi: 10.1097/ICB.0000000000000414. PMID 27617392
- [Background] Raghava S, Hammond M, Kompella UB. Periocular routes for retinal drug delivery. Expert Opin Drug Deliv. 2004 Nov;1(1):99-114. doi: 10.1517/17425247.1.1.99. PMID 16296723
- [Background] Bahar I, Yeung SN, Sella R, Slomovic A. Anterior segment uses of bevacizumab. Curr Opin Ophthalmol. 2012 Jul;23(4):303-16. doi: 10.1097/ICU.0b013e3283548459. PMID 22634640
- [Background] Papadopoulos N, Martin J, Ruan Q, Rafique A, Rosconi MP, Shi E, Pyles EA, Yancopoulos GD, Stahl N, Wiegand SJ. Binding and neutralization of vascular endothelial growth factor (VEGF) and related ligands by VEGF Trap, ranibizumab and bevacizumab. Angiogenesis. 2012 Jun;15(2):171-85. doi: 10.1007/s10456-011-9249-6. PMID 22302382
- [Background] Stewart MW, Rosenfeld PJ. Predicted biological activity of intravitreal VEGF Trap. Br J Ophthalmol. 2008 May;92(5):667-8. doi: 10.1136/bjo.2007.134874. Epub 2008 Mar 20. PMID 18356264
- [Background] Kitchens JW, Do DV, Boyer DS, Thompson D, Gibson A, Saroj N, Vitti R, Berliner AJ, Kaiser PK. Comprehensive Review of Ocular and Systemic Safety Events with Intravitreal Aflibercept Injection in Randomized Controlled Trials. Ophthalmology. 2016 Jul;123(7):1511-20. doi: 10.1016/j.ophtha.2016.02.046. Epub 2016 Apr 12. PMID 27084563